CLINICAL TRIAL: NCT06310239
Title: Osseointegrated Limb Implant Microbiome Population Adaptation Study
Brief Title: Microbiome Population Adaptation Study
Acronym: OLIMPAS
Status: Recruiting | Type: Observational
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: WRNMMC-2023-0434; 67407 (Other Grant/Funding Number: PRORP)
Record Dates: First submitted 2024-02-21; First posted 2024-03-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Amputation With Osseointegration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study subjects: Individuals with a limb amputation who are undergoing an osseointegration surgery
  Interventions: Other: Collection of biologic samples and data

INTERVENTIONS:
Other: Collection of biologic samples and data — * collection of skin flora samples via swabs
  * data collection regarding subject's medications See Detailed Description in Study Description section above for more details

SUMMARY:
The investigators will accomplish our research aims by collecting cutaneous microbiome samples from 50 persons that have undergone the Osseointegration (OI) surgery at eight timepoints, prospectively. The investigators will also collect control samples to correct for turnovers in species compositions that may naturally occur and to compare the residual limb microbiome to the sound contralateral limb. The investigators will sequence the bacterial community using universal bacterial primers. Using these sequences, The investigators will borrow from ecological theory and calculate the alpha and beta diversity. The alpha diversity will determine the species and abundance of each species that are present, while the beata diversity will allow us to compare how species assemblages and frequencies change between time points. Then, the investigators will take a phylogenetic modeling approach to determine if particular species assemblages correlate with rates of wound healing. The investigators will construct phylogenies from the sequences at the different time points and "paint" the rate of wound healing along the phylogeny (e.g., improved, stagnated, worsened). Using Akaike and Bayesian information criterion, the investigators can determine which phylogenetic model best explains the patterns the investigators see across patients. Lastly, the investigators will quantify soft tissue stability and health and correlate this with the homeostasis of the microbial community. Specifically, the investigators will determine if redundant soft tissue leads to altered microbial communities that can impact the rate of wound healing. Finally, the investigators will further stratify these data to compare microbial communities between the sexes, upper versus lower limbs, and proximal versus distal amputations. This work will allow us to better treat infections after OI surgery and can shed light on wound healing process so that the investigators can better treat limb loss patients and the military community as a whole.

DETAILED DESCRIPTION:
Patients that are undergoing to have OI surgery will be asked if they would like to participate in the research study. All the data collected for the study is research related and will be collected on the case report forms ( CRFs) /source documents and will be entered into the Henry Jackson Foundation (HJF) REDCap.

Below is a breakdown of the research-related study procedures. All of these procedures will be done for research purposes, none of them are for the standard of care. The investigators will coincide study visit with clinical visits/ follow ups. The investigators will collect the following information from the patients/clinician:

Baseline/Pre-operative Surgery Stage I

Demographics (DOB, sex, height, weight, BMI, length of residual limb, amputated side, side indicated for surgery, date of amputation, reason for amputation, details of reason for amputation, issues with prior/current prosthesis) Medication: The investigators will collect detailed information about the medications (names, indication, dose, frequency, route. etc.) that the patients are currently taking (including over-the counter medications, vitamins, or herbal treatment).

Hygiene Questionnaire Biome sample (Osseointegrated and control site) Flora Data Collection Sample Questionnaire Flora Data Collection Sample Questionnaire-Control Holger Score System Questionnaire ( It is a score that the investigators is given after they evaluate the participant's skin condition).

Clinical Assessment

Pre-operative Surgery Stage II, Post-Operative 3 Weeks, 3 Months, 6 Months, and 12 Months Follow-Ups from Surgery Stage II

Medication: The patients will be asked about any changes to the medications that they are taking currently.

Hygiene Questionnaire Biome sample (Osseointegrated and control site) Flora Data Collection Sample Questionnaire Flora Data Collection Sample Questionnaire-Control Holger Score System Questionnaire

Post-Operative Surgery Stage II (in the OR)

Flora Data Collection Sample Questionnaire Flora Data Collection Sample Questionnaire-Control Biome sample (Osseointegrated and control site) Holger Score System Questionnaire

24 Months Post-Operative Surgery Stage II

Medication: The patients will be asked about any changes to the medications that they are taking currently.

Hygiene Questionnaire Biome sample (Osseointegrated and control site) Flora Data Collection Sample Questionnaire Flora Data Collection Sample Questionnaire-Control Holger Score System Questionnaire Thighplasty Questionnaire Clinical Assessment

Data collected will include flora samples collections and soft tissue envelop analysis

Flora samples collections

Biome samples will be collected /swabbed by one of the study team members. The swab area of skin or abutment will be about 2 cm x 2 cm.

Samples collecting swabbing sites For unilateral amputation patients Amputated limb: Implant surface, aperture site, the midpoint between amputated site and groin or axillary crease, and amputation site Contralateral limb as a control: as same level as amputated limb (compatible location of swabbing sites to the imputed limb) For the bilateral amputation patients Both amputated limbs: Implant surface, aperture site, the midpoint between amputated site and groin or axillary crease (as control) Anytime a participant has an infection and comes in outside of research-related timepoints The investigators will collect a Biome sample (Osseointegrated and control site), Flora Data Collection Sample Questionnaire, Flora Data Collection Sample Questionnaire-Control, and clinical assessment.

Sample collection swabbing procedures

Flora is the microorganisms that exist in all living things. The investigators will use the swabbing method to collect the participant's skin biome/flora samples on their Osseointegrated and control site. The fresh swab will be in a moistening buffer such as saline or distilled water. One of the study team members will use one hand to stretch the skin site taut. With the other hand, hold the swab so the shaft is parallel to the skin surface. Apply firm pressure and rub the swab back and forth rigorously 50 times (for 30 seconds). The swab will be put in the tube buffer and will be taken to the freezer as soon as possible (within 30 min of collecting). This is a noninvasive procedure that will cause no pain but may cause discomfortable at the collecting site. If the participants ask us to stop to collection the samples because they experience any pain, The investigators will stop to collection the flora samples.

The participant's skin flora samples will be collected at Baseline/Pre-operative Surgery Stage I, Pre-operative Surgery Stage II, Immediate post-operative Surgery Stage II (in the Operation room), Post-Operative 3 Weeks, 3 Months, 6 Months, 12 Months, and 24 months Follow-Ups from Surgery Stage II.

Swab samples processing, storing, and analysis

The swab needs to go in the tube buffer and be taken to the freezer ASAP (within 30 min of collecting). These biome samples will be stored at the -20 º the Surgical Critical Care Initiative (SC2i) freezer located in building#9. Once the investigators have accumulated enough samples, the investigators will send these samples to Zymo Research Corporation for sequencing on dry ice so the samples remain frozen. After the analysis of these samples by Zymo, the results will be sent back as text and a fasta file. The text files will be the results (alpha and beta diversity, species identified, etc.) and the fasta file will be the actual genetic sequence. Zymo will dispose of all unused samples after three months once the study has been completed

The soft tissue envelope analysis

The soft tissue envelope will be measured for redundancy and scored using the Modified Holger Score System. The investigators will document soft tissue redundancy and hypermobility, drainage and irritability, and active infection. Clinical data being collected are demographics (DOB, sex, height, weight, BMI, length of residual limb, amputated side, side indicated for surgery, date of amputation, reason for amputation, details of reason for amputation, issues with prior/current prosthesis), other relevant past and present medical conditions and medications. Questionnaires that will be collected are hygiene (how many times a day do the participants clean participants' residual limb, what product(s) do the participants use to clean their residual limb, do participant apply any product(s), like lotion, after the participants have cleaned their residual limb, if yes what product(s), flora data collection sample questionnaire (date of assessment, flora sample site, flora sample control site, what site collecting from (implant surface, aperture site, contralateral limb) and person collecting sample), Holger Score System (normal skin, reddish, red and moist, granulation tissues and skin complication leading to removal of the abutment, skin overgrowth), Clinical Assessment (soft tissue-redundancy, hypermobility, drainage irritable), wound grade (improved, stagnated and worsened) and thighplasty questionnaire (did the patient have to have a thighplasty).

ELIGIBILITY:
Inclusion Criteria:

* Any adult male or female that will undergo an OI procedure between the ages of 18-75.
* Defense Enrollment Eligibility Reporting System (DEERs) eligible

Exclusion Criteria:

* Inability to provide self-consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female military health care beneficiaries aged 18-75 years old have undergone an osseointegrated percutaneous prosthetic system.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Determine if OI surgery causes changes in the microbiome community using phylogenies | month 36
  We will use phylogenies and phylogenetic comparative methods to quantify the changes in the cutaneous microbiome flora before and after OI surgery. This will be done by comparing phylogenies across time points to determine changes in species lineage composition.
Determine if changes in the microbiome community predicts wound healing using phylogenetic comparative methods | months 36-48
  We will use phylogenetic comparative methods and community turnover rates, quantified via alpha and beta diversity measures, to determine if community perturbations impact wound healing.
Quantify soft tissue health using a modified Holger Score (0 = healthy soft issue and 6 = unhealthy soft tissue) to phylogenetically correlate this with microbiome homeostasis. | months 36-48
  We will clinically quantify soft tissue stability using a modified Holger Score, then, we will use a phylogenetic correlation to determine if soft tissue health drives microbiome homeostasis

SECONDARY OUTCOMES:
Floral profiles | months 40
  We will use phylogenies to build species assemblages profiles (which species are present) for each participant. Then, we will use phylogenetic methods to compare profiles within each patient through time.
Floral colonization | months 42
  We will use the microbial profiles and phylogenies to determine the colonization order of the microbiome after OI surgery by comparing which species are present at baseline and which species are present at the subsequent follow-ups.
Clinical guidelines | month 48
  We will design and write clinical practice guidelines to identify a skin penetration aperture infection and disseminate to the public so others can use the same guidelines
Surgical site questionnaire | month 44
  We will develop and disseminate a questionnaire for the cleaning and maintenance of the skin penetration aperture to correlate hygiene routines and probability of developing a superficial infection.
Post-OI hygiene guidelines | month 46
  We will develop and disseminate a skin penetration aperture hygiene guidelines based on the findings of the microbiome profiles to reduce the probability of developing a superficial infection.
Soft tissue stability guidelines | month 46
  We will develop and disseminate best practice guidelines for clinicians based on our findings to educate surgeons on soft tissue stability and when surgical intervention is needed to correct soft tissue complications.
Holger score validation | Time Frame: month 48
  We will validate our modified Holger Score (0 = healthy soft issue and 6 = unhealthy soft tissue) in osseointegrated patients for the skin penetration aperture by determining the interobserver variation.

CONTACTS AND LOCATIONS:
Overall Officials: Ean R Saberski, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (1):
- Orhopaedic Surgery Service, Walter Reed National Military Medical Center,, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] NIH Human Microbiome Portfolio Analysis Team. A review of 10 years of human microbiome research activities at the US National Institutes of Health, Fiscal Years 2007-2016. Microbiome. 2019 Feb 26;7(1):31. doi: 10.1186/s40168-019-0620-y. PMID 30808411
- [Background] Schmidt BM. Emerging Diabetic Foot Ulcer Microbiome Analysis Using Cutting Edge Technologies. J Diabetes Sci Technol. 2022 Mar;16(2):353-363. doi: 10.1177/1932296821990097. Epub 2021 Feb 12. PMID 33576276
- [Background] Zenga J, Atkinson S, Yen T, Massey B, Stadler M, Bruening J, Peppard W, Reuben M, Hayward M, Mesich B, Buchan B, Ledeboer N, Sanchez JL, Fraser R, Lin CW, Holtz ML, Awan M, Wong SJ, Puram SV, Salzman N. A phase 2 trial of a topical antiseptic bundle in head and neck cancer surgery: Effects on surgical site infection and the oral microbiome. EBioMedicine. 2022 Jul;81:104099. doi: 10.1016/j.ebiom.2022.104099. Epub 2022 Jun 4. PMID 35671624
- [Background] Zeeuwen PL, Boekhorst J, van den Bogaard EH, de Koning HD, van de Kerkhof PM, Saulnier DM, van Swam II, van Hijum SA, Kleerebezem M, Schalkwijk J, Timmerman HM. Microbiome dynamics of human epidermis following skin barrier disruption. Genome Biol. 2012 Nov 15;13(11):R101. doi: 10.1186/gb-2012-13-11-r101. PMID 23153041
- [Background] Xu Z, Hsia HC. The Impact of Microbial Communities on Wound Healing: A Review. Ann Plast Surg. 2018 Jul;81(1):113-123. doi: 10.1097/SAP.0000000000001450. PMID 29746280
- [Background] Dunyach-Remy C, Salipante F, Lavigne JP, Brunaud M, Demattei C, Yahiaoui-Martinez A, Bastide S, Palayer C, Sotto A, Gelis A. Pressure ulcers microbiota dynamics and wound evolution. Sci Rep. 2021 Sep 16;11(1):18506. doi: 10.1038/s41598-021-98073-x. PMID 34531517
- [Background] Wolcott RD, Hanson JD, Rees EJ, Koenig LD, Phillips CD, Wolcott RA, Cox SB, White JS. Analysis of the chronic wound microbiota of 2,963 patients by 16S rDNA pyrosequencing. Wound Repair Regen. 2016 Jan-Feb;24(1):163-74. doi: 10.1111/wrr.12370. Epub 2015 Dec 10. PMID 26463872
- [Background] Gardiner M, Vicaretti M, Sparks J, Bansal S, Bush S, Liu M, Darling A, Harry E, Burke CM. A longitudinal study of the diabetic skin and wound microbiome. PeerJ. 2017 Jul 20;5:e3543. doi: 10.7717/peerj.3543. eCollection 2017. PMID 28740749
- [Background] Loesche M, Gardner SE, Kalan L, Horwinski J, Zheng Q, Hodkinson BP, Tyldsley AS, Franciscus CL, Hillis SL, Mehta S, Margolis DJ, Grice EA. Temporal Stability in Chronic Wound Microbiota Is Associated With Poor Healing. J Invest Dermatol. 2017 Jan;137(1):237-244. doi: 10.1016/j.jid.2016.08.009. Epub 2016 Aug 24. PMID 27566400
- [Background] Gerzina C, Potter E, Haleem AM, Dabash S. The future of the amputees with osseointegration: A systematic review of literature. J Clin Orthop Trauma. 2020 Feb;11(Suppl 1):S142-S148. doi: 10.1016/j.jcot.2019.05.025. Epub 2019 May 31. PMID 31992935
- [Background] Grice EA, Segre JA. The skin microbiome. Nat Rev Microbiol. 2011 Apr;9(4):244-53. doi: 10.1038/nrmicro2537. PMID 21407241
- [Background] Orgel M, Aschoff HH, Sedlacek L, Graulich T, Krettek C, Roth S, Ranker A. Analysis of Stomal Bacterial Colonialization After Transcutaneous Osseointegrated Prosthetic Systems Surgery. JAMA Netw Open. 2022 Jul 1;5(7):e2223383. doi: 10.1001/jamanetworkopen.2022.23383. PMID 35867064
- [Background] Beck JP, Grogan M, Bennett BT, Jeyapalina S, Agarwal J, Bartow-McKenney C, Bugayev J, Kubiak E, Sinclair S, Grice E. Analysis of the Stomal Microbiota of a Percutaneous Osseointegrated Prosthesis: A Longitudinal Prospective Cohort Study. J Orthop Res. 2019 Dec;37(12):2645-2654. doi: 10.1002/jor.24421. Epub 2019 Aug 2. PMID 31317568
- [Background] Branemark R, Berlin O, Hagberg K, Bergh P, Gunterberg B, Rydevik B. A novel osseointegrated percutaneous prosthetic system for the treatment of patients with transfemoral amputation: A prospective study of 51 patients. Bone Joint J. 2014 Jan;96-B(1):106-13. doi: 10.1302/0301-620X.96B1.31905. PMID 24395320
- [Background] Holgers KM, Tjellstrom A, Bjursten LM, Erlandsson BE. Soft tissue reactions around percutaneous implants: a clinical study of soft tissue conditions around skin-penetrating titanium implants for bone-anchored hearing aids. Am J Otol. 1988 Jan;9(1):56-9. PMID 3364537
- [Background] Lenneras M, Tsikandylakis G, Trobos M, Omar O, Vazirisani F, Palmquist A, Berlin O, Branemark R, Thomsen P. The clinical, radiological, microbiological, and molecular profile of the skin-penetration site of transfemoral amputees treated with bone-anchored prostheses. J Biomed Mater Res A. 2017 Feb;105(2):578-589. doi: 10.1002/jbm.a.35935. Epub 2016 Nov 7. PMID 27750392
- [Background] Verbanic S, Shen Y, Lee J, Deacon JM, Chen IA. Microbial predictors of healing and short-term effect of debridement on the microbiome of chronic wounds. NPJ Biofilms Microbiomes. 2020 May 1;6(1):21. doi: 10.1038/s41522-020-0130-5. PMID 32358500
- [Background] Klindworth A, Pruesse E, Schweer T, Peplies J, Quast C, Horn M, Glockner FO. Evaluation of general 16S ribosomal RNA gene PCR primers for classical and next-generation sequencing-based diversity studies. Nucleic Acids Res. 2013 Jan 7;41(1):e1. doi: 10.1093/nar/gks808. Epub 2012 Aug 28. PMID 22933715
- [Background] R Core Team. R: A language and environment for statistical computing. R Foundation for Statistical Computing. 2021. Vienna, Austria. URL https://www.R-project.org/.
- [Background] Grice EA, Kong HH, Conlan S, Deming CB, Davis J, Young AC; NISC Comparative Sequencing Program; Bouffard GG, Blakesley RW, Murray PR, Green ED, Turner ML, Segre JA. Topographical and temporal diversity of the human skin microbiome. Science. 2009 May 29;324(5931):1190-2. doi: 10.1126/science.1171700. PMID 19478181